CLINICAL TRIAL: NCT06228976
Title: A Randomized Controlled Trial Exploring Mindfulness-based Smoking Cessation Intervention Using Mobile Technology in Vietnam
Brief Title: Mindfulness-based, Mobile Health (mHealth) Smoking Cessation Intervention in Vietnam
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanoi University of Public Health (Other)
Collaborators: Georgia State University (Other); National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Hoang Van Minh, Dean, Hanoi University of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: mhealthVN01; 5R01TW010666-05 (NIH)
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Smoking Cessation; Mindfulness; Telemedicine; Smoking
Keywords: smoking cessation; smoking behavior; Mindfulness-based; randomized controlled trial; Vietnam; mobile health
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Arm (Experimental): One or two tailored messages will be sent to participants everyday at designated time for 12 weeks
  Interventions: Behavioral: Mindfulness-based, smoking cessation focused text messages.
- Education Arm (Active Comparator): One tailored message will be sent to participants everyday at designated time for 12 weeks
  Interventions: Behavioral: Educational messages
- Control arm (Active Comparator): One tailored message will be sent to participants everyday at designated time for 12 weeks
  Interventions: Behavioral: Control messages

INTERVENTIONS:
Behavioral: Mindfulness-based, smoking cessation focused text messages. — Participants will receive mindfulness-based, smoking cessation focused text messages everyday for 12 weeks.
  Arms: Intervention Arm
Behavioral: Educational messages — Text messages focus on the health risks of smoking and secondhand smoking, once everyday for 12 weeks.
  Arms: Education Arm
Behavioral: Control messages — Text messages focus on the general healthy lifestyle, once everyday for 12 weeks.
  Arms: Control arm

SUMMARY:
The goals of this a three-arm randomized controlled trial (RCT) is to evaluate the efficacy of mindfulness-based, culturally appropriate, and mobile phone-based smoking cessation intervention among Vietnamese adult male smokers.

The intervention will be delivered via text messages, involving 1,200 adult male smokers, with 400 participants in each of three intervention arms (Cessation Intervention - culturally-adapted smoking cessation messages that incorporate mindfulness; Education Intervention - messages that solely focus on health risks of smoking; Control - basic messages that solely focus on general healthy lifestyle). The investigator will assess cessation rates up to 6-month follow-up, as well as secondary outcomes of knowledge of smoking health risks; stages of change; quit attempts; self-efficacy; cigarettes per day; and nicotine dependence. The investigators hypothesize that participants in the Cessation Intervention group (who will receive culturally-adapted messages) will have higher rates of smoking abstinence, greater knowledge of the health risks of smoking, more transitions from pre-contemplation/contemplation stages to planning/action stages, higher likelihood of making a quit attempt, higher self-efficacy for abstaining from smoking, greater reductions in cigarette consumption, and lower nicotine dependence, compared to participants in the Education Intervention group and Control group.

DETAILED DESCRIPTION:
Cessation Intervention: Participants in the Cessation Intervention group will be divided into two groups (have intention to quit vs. not have intention to quit) based on the participants' stage of change (Transtheoretical Model) [1] at baseline assessment to receive different message libraries during the 12 week intervention. Participants who have intention to quit (at the action or preparation stage of change) will set the quit date at time of enrollment to the study. The two weeks before the quit date, participants will receive 2 messages per day with content focusing on health benefits of quitting, monetary costs of smoking, encouragement and some tips/strategies to prepare for the quit date. Two days around the quit date, participants will receive 3-4 messages per day, and the first five weeks participants will receive 2 messages per day. The content of messages in the first five weeks after the quit date is diverse, providing participants a lot of tips/strategies (including mindfulness practice) to deal with cravings/withdrawal symptoms, benefits of quitting, interactive messages asking the participants' mood and craving levels, motivating messages and encouraging to get supports from family/friends and other smoking cessation resources (i.e., quit line, website). During this period, participants will periodically be asked about maintain smoke-free, and based on the particpants' answer, further messages will provide encouragement to get back on track or stay focus to avoid relapse. From week 6 to week 12, participants will just receive one message per day, with content covers benefits of quitting smoking, motivating messages, tips to avoid cravings/relapse, and interactive messages asking about the participants' smoke free status. Participants who do not have intention to quit will receive messages from another library, with the frequency of one message per day throughout 12 weeks of the intervention. This message library will provide participants knowledge of negative effects of smoking with specific evidences, benefits of quitting, encouraging messages as well as messages to increase the participants self-efficacy in quitting smoking. From week 2 to week 7, participants in this group will receive an interactive message on every 7-day period, asking if the participants want to set a quit date in the next week. If participants answer yes to the question, the participants will be switch to the message library for those who have intention to quit as mentioned above.

Education Intervention Group and Control Group: Participants in the Education Intervention and Control groups will also receive one single message per day for the entire 12-week intervention period. Education Intervention messages will specifically focus on the health risks of smoking and secondhand smoking (i.e., education about health risks, without providing specific strategies for quitting). These messages will be taken from the text message library developed by NCI, and will be directly translated into Chinese and Vietnamese without cultural adaptions. Control messages will provide general health education (not including smoking), including promoting fruit and vegetable intake and low sodium intake; encouraging physical activity; and avoiding drug use/excess alcohol use. These messages will be translated from previous studies that use mHealth approaches to promote healthy lifestyles.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smokers (irrespective of the person's current intention to quit) who are living in the 6 communes in Hai Duong province
* Ability to read and write in Vietnamese
* Ownership of a cell phone and knowledge/ability to send and receive text messages
* Do not have any plan to relocate in the next year
* Agree to receive text messages for 12 weeks
* Agree to be contacted by the research team for follow-ups interviews

Exclusion Criteria:

* Do not agree to participate in the study
* Have serious chronic illnesses or injuries that affect reading and comprehension
* Cannot participate in the intervention activities during the proposed intervention period

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological male
Enrollment: 1200 (Estimated)
Dates: Start 2023-08-27 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence smoking abstinence | At 12 weeks, at 16 weeks and 36 weeks
  Whether the participant smoked cigarette at all, even a puff, in the last 7 days
30-day point prevalence smoking abstinence | At 12 weeks, at 16 weeks and 36 weeks
  Whether the participant smoked cigarette at all, even a puff, in the last 30 days

SECONDARY OUTCOMES:
Knowledge about health risks of smoking and secondhand smoking | At 12 weeks, at 16 weeks and 36 weeks
  The participants will answer whether smoking caused certain diseases or not.
Stage of change | At 12 weeks, at 16 weeks and 36 week
  The participants will be asked about readiness to quit smoking, and when do the participants plan to quit smoking.
Quit attempts within the last 30 days | At 12 weeks, at 16 weeks and 36 weeks
  Number of quit attempts made that last longer than 01 day because the participant want to quit smoking. The duration of the longest quit attempt made in the last 30 days.
Self-efficacy for abstaining from smoking | At 12 weeks, at 16 weeks and 36 weeks
  The participant will be asked about abstaining from smoking in positive affect/social, negative affect, and habitual/craving situations
Number of cigarettes smoked per day | At 12 weeks, at 16 weeks and 36 weeks
  The participants will be asked about number of cigarettes smoked per day
Nicotine dependency | At 12 weeks, at 16 weeks and 36 weeks
  The participant's nicotine dependency will be assessed using the Fagerstrom Test for Nicotine Dependence

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi University of Public Health, Hanoi, Vietnam

DOCUMENTS (1):
  • Informed Consent Form (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT06228976/ICF_000.pdf